CLINICAL TRIAL: NCT00933439
Title: Assessment of Cognitive Functioning Before and After Treatment With Duloxetine
Acronym: DULOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Prabha Sunderajan, Clinical Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Duloxetine
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder; Cognitive Function; Psychosocial Function
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Approximately 30 participants with major depressive disorder and concentration and/or cognition difficulties, recruited from the community and physician referrals, will be treated with duloxetine for 12 weeks. Their cognitive performance will be assessed pre- and post-treatment with a cognitive testing battery.

SUMMARY:
The purpose of this study is to study the effect of duloxetine treatment on (1) cognitive functions, the brain mechanisms involved with thinking, reasoning, learning, and remembering; (2) psychosocial functions, how someone interacts with his/her social environment; and (3) the relationship between these two functions, in people who have major depressive disorder, a severe form of depression.

DETAILED DESCRIPTION:
People who have difficulties with concentration and/or cognition as part of their depression will be treated with duloxetine for 12 weeks and their cognitive performance will be assessed before and after treatment using cognitive tests. Eligible participants will have eight clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent
* Primary diagnosis of Major Depressive Disorder (MDD)
* Age 18-45
* Screening and baseline Hamilton Rating Scale for Depression (HRSD) 17-item score greater than or equal to 16 or Clinical Global Impression (CGI) score of at least 4
* Subjective report of difficulties with cognition and/or concentration and score of 2 or greater on the Inventory for Depressive Symptomatology (IDS-C(30)) item addressing this symptom (#16: Concentration and Decision Making)

Exclusion Criteria:

* Presence of significant comorbid condition based on laboratory tests, physician information, or evidence at examination
* Patient report or evidence (based on physical examination or laboratory tests) of existing liver disease
* Presence of other psychological disorders, including depression due to other comorbid conditions, currently suicidal or high suicide risk, current or past psychotic disorders of any type, bipolar disorder (I, II, or NOS), schizophrenia, or schizoaffective disorder, anorexia, bulimia, obsessive compulsive disorder, alcohol or substance abuse within the last 6 months, or patients with comorbid psychiatric conditions that are relative or absolute contraindications to the use of duloxetine
* Concomitant pharmacological or psychotherapeutic treatment including but not limited to antidepressants, anxiolytics, neuroleptics, mood stabilizers, and/or other agents without proven antidepressant efficacy, cognitive behavioral therapy; current use of other medications that would be contraindicated with duloxetine, as determined by the study doctor
* Hospitalization for mental illness within the past year
* Not fluent in spoken and written English
* For women, currently pregnant, planning to become pregnant in the next year, or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 8 weeks

SECONDARY OUTCOMES:
Psychosocial function | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prabha Sunderajan, MD, Principal Investigator — UT Southwestern Medical Center - Department of Psychiatry
Locations (1):
- Mood Disorders Research Program and Clinic - UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Greer TL, Sunderajan P, Grannemann BD, Kurian BT, Trivedi MH. Does duloxetine improve cognitive function independently of its antidepressant effect in patients with major depressive disorder and subjective reports of cognitive dysfunction? Depress Res Treat. 2014;2014:627863. doi: 10.1155/2014/627863. Epub 2014 Jan 19. PMID 24563781